CLINICAL TRIAL: NCT04788043
Title: A Phase 2 Study of Magrolimab and Pembrolizumab in Relapsed or Refractory Classic Hodgkin Lymphoma
Brief Title: Study of Magrolimab and Pembrolizumab in Relapsed or Refractory Classic Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-56995; LYMHD0019 (Other: OnCore); NCI-2022-05298 (Registry Identifier: NCI- Clinical Trials Reporting Program)
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Hodgkin Lymphoma; Classic Hodgkin Lymphoma; Relapsed Classical Hodgkin Lymphoma; Refractory Classic Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — magrolimab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Magrolimab (Hu5F9 G4) and pembrolizumab (Experimental): All subjects will have a baseline PET CT and excisional or core needle biopsy within 1 month of study enrollment and baseline electrocardiogram and laboratory studies within 1 week of study enrollment. All subjects will receive treatment with magrolimab and pembrolizumab according to the dosing schedule. Magrolimab IV given on cycle 1, 2 and 3. Pembrolizumab 200 mg IV given on Cycle 1, 2 and 3. Patients may continue to receive treatment on the study for a maximum of 24 months or until progression of disease, unacceptable toxicity, or bridge to stem cell transplantation (SCT).
  Interventions: Drug: Magrolimab; Drug: Pembrolizumab; Procedure: PET/CT

INTERVENTIONS:
Drug: Magrolimab — 45 mg/kg with dose escalation starting at 1 mg/kg IV Infusion
  Other Names: Hu5F9-G4; ONO-7913; anti-CD47 monoclonal antibody Hu5F9-G4
Drug: Pembrolizumab — 200 mg IV infusion
  Other Names: Keytruda; MK-3475; SCH 900475; anti-PD-1 monoclonal antibody MK-3475
Procedure: PET/CT — Scan
  Other Names: Positron Emission Tomography - Computed Tomography (PET/CT)

SUMMARY:
The purpose of this study is to test the safety and efficacy of magrolimab in combination with pembrolizumab in patients with Hodgkin lymphoma.

DETAILED DESCRIPTION:
Primary Objectives:

- To assess the complete remission (CR) rate of magrolimab in combination with pembrolizumab in adult subjects with relapsed or refractory cHL

Secondary Objectives:

* To assess the safety and tolerability of magrolimab in combination with pembrolizumab in adult subjects with relapsed or refractory cHL
* To assess the overall response rate (ORR)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Biopsy proven relapsed or refractory cHL
* Prior treatment with at least two systemic therapies
* Metabolically active measurable disease by PET imaging per the 2014 Lugano criteria
* Hemoglobin ≥ 9.5 g/dL
* Absolute neutrophil count ≥ 1,000 cells/μL without G-CSF support within 3 weeks prior to enrollment
* Platelet count ≥ 75,000 cells/μL
* Creatinine clearance > 40 mL/min per the Cockroft-Gault formula
* Total bilirubin < 1.5 x upper limit of normal (ULN) (or < 3.0 x ULN and primarily unconjugated in subjects with a history of Gilbert's syndrome)
* Negative urine or serum pregnancy test within 30 days of enrollment and within 72 hours before the first administration of magrolimab for women of childbearing potential
* Women of childbearing potential must be willing to use at least 1 highly effective method of contraception during the study and continue for 4 months after the last dose of magrolimab
* Male subjects who are sexually active with a woman of childbearing potential and who have not had vasectomies must be willing to use a barrier method of contraception during the study and for 4 months after the last dose of magrolimab
* Ability to understand and the willingness to sign the written IRB approved informed consent document
* Must be willing and able to comply with the clinic visits and procedures outlined in the study protocol

Exclusion Criteria:

* Prior treatment with a PD-1 inhibitor within 3 months prior to enrollment
* Prior treatment with antibodies targeting CD47 or SIRPα2
* Prior allogeneic hematopoietic cell transplantation
* Systemic autoimmune disorder on chronic immunosuppression (defined as ≥ 10 mg of prednisone daily)
* RBC transfusion dependence, defined as requiring more than 2 units of RBCs during the 4-week period prior to screening
* History of hemolytic anemia, autoimmune thrombocytopenia, or Evan's syndrome within the last 3 months
* Second malignancy not in complete remission for at least 1 year, excluding fully resected non melanoma skin cancer or localized prostate cancer
* Women who are pregnant or breast feeding
* HIV or hepatitis B or C infection with active viral replication by PCR
* Second malignancy not in complete remission for at least 1 year, excluding fully resected non-melanoma skin cancer or localized prostate cancer
* Active cardiac disease including unstable angina, decompensated congestive heart failure, or severe uncontrolled conduction abnormalities
* History of non-infectious pneumonitis requiring corticosteroids or current pneumonitis
* Significant medical conditions, as assessed by the investigators and IND holder, that would substantially increase the risk benefit ratio of participating in the study
* History of psychiatric illness or substance abuse likely to interfere with ability to comply with protocol requirements
* Received a live or live attenuated vaccine within 30 days before the first dose of study intervention
* Received any anti-cancer therapy within 2 weeks prior to the first dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) | 2 years
  Each participant's response to treatment will be assessed per the Lugano criteria. The criteria are:
  * Complete Response (CR): Complete disappearance of all lesions, evidence, and effects of disease
  * Partial Response (PR): ≥50% decrease in SPD of the 6 largest lesions with no increase in the size of the other nodes; splenic / hepatic nodules regress ≥50%, and with no new sites of disease
  * Stable disease (SD): less than PR.
  * Progressive disease (PD): sum of the product of dimensions (SPD) of lesions increased ≥50% from smallest value The outcome will be reported as the number of participants with a CR after 4 and 8 cycles of treatment (4 and 8 months), and if CR is achieved anytime within 2 years ("overall").

SECONDARY OUTCOMES:
Magrolimab related Adverse Events | 4 months
  Magrolimab safety and tolerability will be assessed on the basis of magrolimab related adverse events occurring within 4 cycles of treatment (4 months). The outcome will be reported as the number of magrolimab related adverse events judged mild (Grade 1), moderate (Grade 2), severe (Grade 3), life threatening (Grade 4), or fatal (Grade 5), numbers without dispersion.

OTHER OUTCOMES:
Overall Response (OR) | 8 months
  Overall response (OR) is defined as the sum of participants who achieve a complete response (CR) plus the number of participants who achieve a partial response (PR). Treatment response will be assessed per the Lugano criteria (aka the Cheson criteria). The criteria are:
  * CR: Complete disappearance of all lesions, evidence, and effects of disease
  * PR: ≥50% decrease in SPD of the 6 largest lesions with no increase in the size of the other nodes; splenic / hepatic nodules regress ≥50%, and with no new sites of disease
  * Stable disease (SD): less than PR.
  * Progressive disease (PD): sum of the product of dimensions (SPD) of lesions increased ≥50% from smallest value The outcome will be reported as the number of participants with either a CR or a PR after 4 and 8 cycles of treatment (4 and 8 months). For participants who undergo a subsequent stem cell transplant, the value will be recorded as the time to transplant (censored).

CONTACTS AND LOCATIONS:
Overall Officials: Ranjana H Advani, MD, Principal Investigator — Stanford Universiy
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No